CLINICAL TRIAL: NCT05368259
Title: A Prospective, Open-Label, Multi-Center, Randomized, Pivotal Safety and Efficacy Study of the Allurion Gastric Balloon System + Moderate Intensity Lifestyle Modification Therapy Program vs. Moderate Intensity Lifestyle Modification Therapy Program for the Treatment of Adults With Obesity
Brief Title: The AUDACITY Study (AllUrion Device in Adults With Clinical ObesITY)
Acronym: AUDACITY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allurion Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRL-1000-0007
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AGBS + Moderate Intensity Lifestyle Therapy Group (Experimental): Patients randomized to treatment will receive the AGBS device
  Interventions: Device: AGBS
- Moderate Intensity Lifestyle Therapy (CONTROL) Group (No Intervention): Patients randomized to the control arm will receive moderate-intensity lifestyle therapy.

INTERVENTIONS:
Device: AGBS — The AGBS is designed to promote weight loss in individuals with obesity. The AGBS includes the Allurion Balloon, which is a temporary gastric balloon that promotes weight loss in individuals with obesity. The AGBS consists of up to 2 balloons placed during a 1-year period.
  Other Names: Allurion Gastric Balloon System (AGBS)
  Arms: AGBS + Moderate Intensity Lifestyle Therapy Group

SUMMARY:
The objective for this clinical study is to provide FDA with clinical evidence regarding the effectiveness and safety of the AGBS + moderate intensity lifestyle modification therapy program, indwell time of the AGBS inside the stomach, and outcomes at 48 weeks.

DETAILED DESCRIPTION:
Prospective, open-label, multi-center, randomized study comparing the AGBS + moderate intensity lifestyle modification therapy program vs. moderate intensity lifestyle modification therapy program for the treatment of adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years and ≤ 65 years of age
2. BMI ≥30 kg/m2 and ≤ 40 kg/m2
3. Have signed study-specific Informed Consent Form
4. Willing to comply with study requirements, including follow-up visits
5. Documented negative pregnancy test in women of childbearing potential
6. Women of childbearing potential not intending to become pregnant for the duration of study participation. (Note: Women of childbearing potential must not be nursing at the time of treatment).
7. Fully ambulatory without any severe chronic orthopedic disease that requires reliance on crutches, walkers, or a wheelchair that could preclude exercise during the study
8. At least one unsuccessful attempt at weight loss, such as self-administered, commercial, or medically supervised lifestyle therapy program attempted within the 24 months preceding enrollment

Exclusion Criteria:

1. Unable to walk 400 meters (the length of one loop of a track and field race track) without the use of an assistance device (e.g. cane, crutches, walker, wheel chair)
2. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease
3. Pre-existing significant respiratory disease such as chronic obstructive pulmonary disease (COPD), severe sleep apnea and pneumonia
4. Previous bariatric surgery including adjustable gastric band and endoscopic sleeve gastroplasty, or likely to undergo bariatric surgery during the study period
5. Previous use of an intragastric gastric balloon
6. Current use of an intragastric device, PlenityTM and digital weight loss solutions (e.g. Noom or Calibrate)
7. History of any cancer other than non-melanoma skin cancer or papillary thyroid cancer within the last 5 years
8. Benign or malignant gastrointestinal tumors
9. History of chronic pancreatitis or acute pancreatitis within 12 months of enrollment
10. History of, or current, small bowel obstruction
11. History of severe GI motility disorder, such as severe gastroparesis
12. History of any esophageal, gastric, or small bowel surgery
13. History of, or current inflammatory bowel disease
14. Any history of intraperitoneal adhesions
15. Any history of open abdominal or gynecological surgery and/or radiation therapy to the abdomen, with the exception of cesarean sections performed at least 12 months prior to study enrollment
16. History of/or signs and symptoms of/or radiographic evidence of esophageal, gastric, or duodenal disease including, but not limited to hiatal hernia ≥5cm, inflammatory diseases, varices, severe gastroparesis, recent history of gastric or duodenal ulcers, stricture/stenosis, achalasia, severe GERD requiring maximal medical therapy, or LA Grade B, C, or D esophagitis
17. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma)
18. Immunocompromised due to medications or medical disease or diagnosed with HIV
19. History of genetic or endocrine causes of obesity not adequately controlled by medication, including hypothyroidism
20. Type 1 diabetes or Type 2 diabetes with HgbA1c ≥ 7%, or treated with any anti-diabetic medications other than metformin
21. Significant acute and/or chronic infections
22. Severe coagulopathy defined as INR 1.5 or higher or platelet count <150, hepatic insufficiency, or cirrhosis
23. Unable or unwilling to discontinue use of aspirin and/or nonsteroidal anti-inflammatory agents (NSAIDs) at least 7 days prior to Allurion Deployment and continuing for 7 days after the Allurion Balloon is excreted
24. Currently taking the following medications (within 30 days prior to enrollment) and/or there is a need or anticipated need for these medications during the study: Excluded Medications Systemic corticosteroids Anticoagulant therapy (e.g., warfarin, dabigatran) or anti-platelet therapy Immunosuppressive therapy (e.g., azathioprine, cyclosporine) Narcotics, opiates, or benzodiazepines Insulin for treatment of diabetes Anti-seizure therapy (e.g., clonazepam, phenytoin) Anti-arrhythmics (e.g., amiodarone)
25. Inability or unwillingness to take anti-emetics during the device residence
26. Prescription or over-the- counter weight loss medication known to cause significant weight gain or weight loss within 90 days of study enrollment through study participation
27. Uncontrolled or severe psychiatric disease other than mild depression with a patient health questionnaire score of 9 or below
28. History of pulmonary embolism or deep venous thrombosis
29. Has cardiac pacemaker or other electric implantable device
30. Anemia defined as either:

    Hgb <11 g/dL for females, <12 g/dL for males
31. Cessation of any nicotine product within 3 months of enrollment or plans to quit use during the study
32. Documented total body weight loss of ≥ 5% anytime 6 months preceding enrollment
33. Residing in a location without access to study site medical resources
34. History of or currently active eating disorders including night eating syndrome (NES), bulimia, or binge eating disorder
35. Unwilling to refrain from any reconstructive and/or cosmetic surgery that may affect body weight during the study such as mammoplasty and lipoplasty
36. Current, or history of, illicit drug use (defined per state law) or excessive alcohol use
37. Enrolled in another investigational study that has not completed the required primary endpoint follow-up period (Note: Subjects involved in a long-term surveillance phase of another study are eligible for enrollment in this study).
38. Current Use (within the last month) of any smoked or non-smoked marijuana products that contain THC or unwilling to abstain from THC containing marijuana products during the trial.
39. Any conditions that, in the opinion of each site investigator, may render the subject unable to complete the study with a likely final outcome, or lead to difficulties for subject compliance with study requirements, or could confound study data.
40. Subject is not of sufficient medical health as determined by the Investigator to participate in the study.
41. Employees/family members of Allurion Technologies or any of its affiliates or contractors
42. Immediate employees/family members of the Investigator, sub- Investigators, or their medical office or practice, or surgical, bariatric or hospital organizations at which study procedures may be performed
43. An immediate family member (by marriage or blood relationship) of another subject already enrolled in the study
44. Positive breath or stool test for H. Pylori
45. History of covid-19 with any residual symptoms
46. Known or suspected allergies to polyurethane
47. Uncontrolled high blood pressure defined as ≥160/100 mmHg with or without medications
48. Uncontrolled high cholesterol or triglycerides defined as LDL ≥190 mg/dL or triglycerides ≥500 mg/dL
49. Inability to swallow Allurion Practice Capsule

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Responder Rate (RR) dichotomized at 5% TBWL at 48 week | 48 weeks
  Responder Rate (RR) dichotomized at 5% TBWL at 48 weeks is significantly greater than 50%
%TBWL is significantly greater than Control Group mean %TBWL at 48 weeks | 48 weeks
  %TBWL is significantly greater than Control Group mean %TBWL at 48 weeks, with a super superiority margin of 3.0%

SECONDARY OUTCOMES:
Responder Rate (RR) dichotomized at both 5% and 10% TBWL at both 16 and 24 weeks | 48 weeks
  Responder Rate (RR) dichotomized at both 5% and 10% TBWL at both 16 and 24 weeks: RR per treatment will be assessed using an exact binomial test and compared between treatments using a two-sided Fisher Exact test; p-values will be descriptive statistics.

OTHER OUTCOMES:
RR dichotomized at 10% TBWL at both 40 and 48 weeks | 48 Weeks
  Among those receiving a second balloon, RR dichotomized at 10% TBWL at both 40 and 48 weeks: RR per treatment will be assessed using an exact binomial test and compared between treatments using a two-sided Fisher Exact test; p-values will be descriptive statistics.
Change in body fatness as measured by Body Mass Index (BMI) at 24 and 48 weeks | 48 Weeks
  Change in BMI (kg/m2) will be calculated as: BMI at follow-up - Baseline BMI Change in BMI will be assessed using a paired t-test within each treatment group and compared between treatments using a two-group unpaired t-test; p-values will be descriptive statistics.
Change in metabolic parameters | 48 Weeks
  Change from screening/baseline in metabolic parameters at 48 weeks. These include HbA1c, total cholesterol, HDL-C, LDL-C, Triglycerides and LFTs. Change in metabolic parameters will be assessed using a paired t-test within each treatment group and compared between treatments using a two-group unpaired t-test; p-values will be descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars-Sinai, Los Angeles, California
  - University of Colorado, Anschutz Health and Wellness Center, Aurora, Colorado
  - University of Miami, Miller School of Medicine, Doral, Florida
  - Chicago Institue of Advanced Surgery, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Luke's Hospital Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health, New Hyde Park, New York
  - Atrium Health Care, Charlotte, North Carolina
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Center for Surgical Weight Loss, Nashville, Tennessee
  - UT Health Science Center at Houston, Bellaire, Texas
  - Segar MD, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided